CLINICAL TRIAL: NCT01519479
Title: An Examination of Palliative Care as Standard Practice for Heart Failure Patients
Brief Title: Palliative Care for Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allina Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 3601-2
Record Dates: First submitted 2012-01-19; First posted 2012-01-27 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Heart Failure
Keywords: Congestive Heart Failure; Heart Failure; Palliative Care; Palliative Medicine
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Palliative Care Consultation (Experimental): Participant will get one palliative care consultation while in the hospital. The participants desire for subsequent palliative care visits will be determined and mutually agreed upon at the initial consultation.
  Interventions: Other: Palliative Care Consultation
- Control (Active Comparator): Usual care for HF patient which may include a palliative care consult if ordered by treating physician.
  Interventions: Other: Control

INTERVENTIONS:
Other: Palliative Care Consultation — Intervention patient would receive an inpatient palliative care consultation to focus on comprehensive symptom assessment, create goals of care/treatment plan which include recommendations and referrals.
  Other Names: palliative care consults; palliative care medicine
  Arms: Palliative Care Consultation
Other: Control — The control group would receive usual care and could receive a palliative consult if ordered by the treating provider
  Other Names: palliative care consult; palliative care medicine
  Arms: Control

SUMMARY:
The purpose of this study is to assess the impact of palliative care consultation on quality of life and symptom management for patients hospitalized with acute heart failure with a randomized control trial at Abbott Northwestern Hospital.

DETAILED DESCRIPTION:
Research questions:

Q1. Does the provision of palliative care to heart failure patients yield higher quality of life, increased symptom management, or reduced depression compared to heart failure patients not receiving palliative care?

Q2. Does the provision of palliative care to heart failure patients result in differential use of medical services (lower hospital days and readmission) compared to heart failure patients not receiving systematic palliative care?

ELIGIBILITY:
Inclusion Criteria:

* Abbott Northwestern Hospital inpatient adults with a diagnosis of acute heart failure

Exclusion Criteria:

* Are not an inpatient at Abbott Northwestern Hospital
* Are in the ICU
* On a ventilator
* Are pre-or post heart transplant
* Have a ventricular assist device (VAD)
* Determined to be actively dying
* Have cognitive impairments such that informed consent would not be possible,
* Are not proficient in the English language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2012-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Is there an impact on quality of life with the addition of palliative care intervention? | Change from baseline in quality of life score at 3 months
  Assessment Tools:
  *Quality of Life-Minnesota Living with Heart Failure questionnaire (MLHF)

SECONDARY OUTCOMES:
Differential use of medical services- 30 day readmission | 30 Days
  *Number of readmissions in 30 days of discharge from initial enrollment hospitalization.
Is there an impact on Symptom Severity with the addition of palliative care | Change from baseline in symptom severity score at 3 months
  Assessment tool:
  *Symptom Severity - Edmonton Symptom Assessment scale (ESAS)
Is there an impact on depression with the addition of palliative care intervention? | Change from baseline in depression score at 3 months
  Assessment Tool:
  *Depression- Patient Health Questionnaire (PHQ-9)

CONTACTS AND LOCATIONS:
Overall Officials: Justin Kirven, MD, Principal Investigator — Allina Health System
Locations (1):
- Abbott Northwestern Hospital, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Bakitas M, Lyons KD, Hegel MT, Balan S, Brokaw FC, Seville J, Hull JG, Li Z, Tosteson TD, Byock IR, Ahles TA. Effects of a palliative care intervention on clinical outcomes in patients with advanced cancer: the Project ENABLE II randomized controlled trial. JAMA. 2009 Aug 19;302(7):741-9. doi: 10.1001/jama.2009.1198. PMID 19690306
- [Background] Temel JS, Greer JA, Muzikansky A, Gallagher ER, Admane S, Jackson VA, Dahlin CM, Blinderman CD, Jacobsen J, Pirl WF, Billings JA, Lynch TJ. Early palliative care for patients with metastatic non-small-cell lung cancer. N Engl J Med. 2010 Aug 19;363(8):733-42. doi: 10.1056/NEJMoa1000678. PMID 20818875
- [Background] Smith ER. Heart failure--are we making progress? Can J Cardiol. 2002 Oct;18(10):1124-5. No abstract available. PMID 12420047
- [Background] Morrison RS, Dietrich J, Ladwig S, Quill T, Sacco J, Tangeman J, Meier DE. Palliative care consultation teams cut hospital costs for Medicaid beneficiaries. Health Aff (Millwood). 2011 Mar;30(3):454-63. doi: 10.1377/hlthaff.2010.0929. PMID 21383364
- [Background] Jovicic A, Holroyd-Leduc JM, Straus SE. Effects of self-management intervention on health outcomes of patients with heart failure: a systematic review of randomized controlled trials. BMC Cardiovasc Disord. 2006 Nov 2;6:43. doi: 10.1186/1471-2261-6-43. PMID 17081306
- [Background] Wilson E. Congestive heart failure: A national priority. Can J Cardiol. 2001 Dec;17(12):1243-4. No abstract available. English, French. PMID 11773934
- [Background] Wolinsky FD, Overhage JM, Stump TE, Lubitz RM, Smith DM. The risk of hospitalization for congestive heart failure among older adults. Med Care. 1997 Oct;35(10):1031-43. doi: 10.1097/00005650-199710000-00005. PMID 9338529
- [Background] Roger VL, Weston SA, Redfield MM, Hellermann-Homan JP, Killian J, Yawn BP, Jacobsen SJ. Trends in heart failure incidence and survival in a community-based population. JAMA. 2004 Jul 21;292(3):344-50. doi: 10.1001/jama.292.3.344. PMID 15265849
- [Background] Stuart B. Palliative care and hospice in advanced heart failure. J Palliat Med. 2007 Feb;10(1):210-28. doi: 10.1089/jpm.2006.9988. PMID 17298270
- [Background] Goodlin SJ. Palliative care in congestive heart failure. J Am Coll Cardiol. 2009 Jul 28;54(5):386-96. doi: 10.1016/j.jacc.2009.02.078. PMID 19628112
- [Background] Stewart S, MacIntyre K, Hole DJ, Capewell S, McMurray JJ. More 'malignant' than cancer? Five-year survival following a first admission for heart failure. Eur J Heart Fail. 2001 Jun;3(3):315-22. doi: 10.1016/s1388-9842(00)00141-0. PMID 11378002
- [Background] Enguidanos SM, Cherin D, Brumley R. Home-based palliative care study: site of death, and costs of medical care for patients with congestive heart failure, chronic obstructive pulmonary disease, and cancer. J Soc Work End Life Palliat Care. 2005;1(3):37-56. doi: 10.1300/J457v01n03_04. PMID 17387068
- [Background] Rabow MW, Dibble SL, Pantilat SZ, McPhee SJ. The comprehensive care team: a controlled trial of outpatient palliative medicine consultation. Arch Intern Med. 2004 Jan 12;164(1):83-91. doi: 10.1001/archinte.164.1.83. PMID 14718327
- [Background] Archana R, Gray D. The quality of life in chronic disease--heart failure is as bad as it gets. Eur Heart J. 2002 Dec;23(23):1806-8. doi: 10.1053/euhj.2002.3309. No abstract available. PMID 12445531
- [Background] O'Connor CM, Joynt KE. Depression: are we ignoring an important comorbidity in heart failure? J Am Coll Cardiol. 2004 May 5;43(9):1550-2. doi: 10.1016/j.jacc.2004.02.003. No abstract available. PMID 15120810
- [Background] Gottlieb SS, Khatta M, Friedmann E, Einbinder L, Katzen S, Baker B, Marshall J, Minshall S, Robinson S, Fisher ML, Potenza M, Sigler B, Baldwin C, Thomas SA. The influence of age, gender, and race on the prevalence of depression in heart failure patients. J Am Coll Cardiol. 2004 May 5;43(9):1542-9. doi: 10.1016/j.jacc.2003.10.064. PMID 15120809
- [Background] Albert NM, Fonarow GC, Abraham WT, Gheorghiade M, Greenberg BH, Nunez E, O'Connor CM, Stough WG, Yancy CW, Young JB. Depression and clinical outcomes in heart failure: an OPTIMIZE-HF analysis. Am J Med. 2009 Apr;122(4):366-73. doi: 10.1016/j.amjmed.2008.09.046. PMID 19332232
- [Background] Rector TS, Cohn JN. Assessment of patient outcome with the Minnesota Living with Heart Failure questionnaire: reliability and validity during a randomized, double-blind, placebo-controlled trial of pimobendan. Pimobendan Multicenter Research Group. Am Heart J. 1992 Oct;124(4):1017-25. doi: 10.1016/0002-8703(92)90986-6. PMID 1529875
- [Background] Rector TS, Kubo SH, Cohn JN. Validity of the Minnesota Living with Heart Failure questionnaire as a measure of therapeutic response to enalapril or placebo. Am J Cardiol. 1993 May 1;71(12):1106-7. doi: 10.1016/0002-9149(93)90582-w. No abstract available. PMID 8475878
- [Background] Rector, T.S., Overview of The Minnesota Living with Heart Failure Questionnaire. 2005, University of Minnesota.
- [Background] Chang VT, Hwang SS, Feuerman M. Validation of the Edmonton Symptom Assessment Scale. Cancer. 2000 May 1;88(9):2164-71. doi: 10.1002/(sici)1097-0142(20000501)88:93.0.co;2-5. PMID 10813730
- [Background] Nekolaichuk C, Watanabe S, Beaumont C. The Edmonton Symptom Assessment System: a 15-year retrospective review of validation studies (1991--2006). Palliat Med. 2008 Mar;22(2):111-22. doi: 10.1177/0269216307087659. PMID 18372376
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Peters-Klimm F, Campbell S, Muller-Tasch T, Schellberg D, Gelbrich G, Herzog W, Szecsenyi J. Primary care-based multifaceted, interdisciplinary medical educational intervention for patients with systolic heart failure: lessons learned from a cluster randomised controlled trial. Trials. 2009 Aug 13;10:68. doi: 10.1186/1745-6215-10-68. PMID 19678944
- [Background] Peters-Klimm F, Kunz CU, Laux G, Szecsenyi J, Muller-Tasch T. Patient- and provider-related determinants of generic and specific health-related quality of life of patients with chronic systolic heart failure in primary care: a cross-sectional study. Health Qual Life Outcomes. 2010 Sep 13;8:98. doi: 10.1186/1477-7525-8-98. PMID 20831837
- [Background] McCarthy M, Lay M, Addington-Hall J. Dying from heart disease. J R Coll Physicians Lond. 1996 Jul-Aug;30(4):325-8. PMID 8875378
- [Result] Sidebottom AC, Jorgenson A, Richards H, Kirven J, Sillah A. Inpatient palliative care for patients with acute heart failure: outcomes from a randomized trial. J Palliat Med. 2015 Feb;18(2):134-42. doi: 10.1089/jpm.2014.0192. Epub 2014 Dec 5. PMID 25479182